CLINICAL TRIAL: NCT03489408
Title: Post-Approval Prospective Study - Conventus CAGE™ PH for Use in Proximal Humerus Fracture Fixation - Study ID 5807
Brief Title: Post-Approval Prospective Study - Conventus CAGE™ PH for Use in Proximal Humerus Fracture Fixation
Status: Terminated | Type: Observational
Why Stopped: Study stopped due to business decision to not continue to gather clinical evidence on product
Sponsor: Conventus Orthopaedics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 5807
Record Dates: First submitted 2018-02-16; First posted 2018-04-05 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-01

CONDITIONS: Humeral Fractures, Proximal
Keywords: Proximal humerus fracture fixation; trauma
MeSH Terms: conditions — Shoulder Fractures; Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Conventus Cage™ PH — Proximal humeral fracture fixation

SUMMARY:
The purpose of this study is to collect device and procedure experience in everyday clinical practice. The patients are being asked to participate in this study because they are a surgical candidate for the treatment of a broken shoulder and are considering treatment with the PH Cage device.

DETAILED DESCRIPTION:
The Conventus CAGE™ PH (PH Cage) System Post-Approval Prospective Study (Study) is a multi-center, prospective, post-approval clinical study designed to collect device and procedure experience in everyday clinical practice.

Specifically, the study will provide:

1. Device safety and patient outcome data.
2. Device usage data.
3. Performance data for the implant procedure.
4. Publications.
5. Early economic benefit data.

Patient Assessments Demographic and general health data will be collected on all patients at the baseline appointment to ensure subjects meet inclusion/exclusion criteria. In addition, to these data, x-rays and adverse event reports related to the implanted device, surgical procedure and/or study data collection methods will be collected.

Patients will be seen at baseline, 2-, 6- and 12-week, 1- and 2-year post op.

Patient participation in this study is voluntary. However, post-implant patient follow-up adds to the medical community's understanding of proximal humerus fracture patient outcomes, as well as the safety and performance of the PH Cage.

ELIGIBILITY:
Inclusion Criteria:

The following criteria, in accordance with the product labelling (Instructions For Use), should be considered when selecting patients for inclusion in this Study:

* Patient must be of at least legal age of consent according to applicable State Law.
* Patient is able to understand and provide written consent.
* Patient is willing and able to cooperate with post-operative instructions, including follow-up examinations and limitations of strenuous activities involving the injured extremity.

Exclusion Criteria:

* The PH Cage should not be implanted in patients with suspected or known allergies to titanium or nickel.
* Patients with open wound fractures.
* Patients with ipsilateral injures or concomitant operation(s) that will have a material impact on the study. Such injuries/ operations are those that affect general health status or the function of the injured extremity.
* Pregnant patients.
* Patients with current or history of mental illness and/or dementia.
* Patients with current or history of alcoholism and/or chemical substance abuse.
* Patient has a medical condition(s) that precludes cooperation with the rehabilitation regimen.
* Patient has active infection at the operative site or other active systemic infection.
* Patient has a pathologic proximal humerus fracture.
* Patients proximal humerus fracture extends into the diaphysis.
* Patient has associated glenohumeral dislocation.
* Patient has ipsilateral injury or concomitant surgery that will have a material impact on the study, such that the injury/surgery affects the patients' health status or the function of the injured extremity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is a prospective, single arm study of patients who are indicated for and have received an FDA cleared Conventus PH Cage.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-02-17 (Actual); Study Completion 2020-02-17 (Actual)

PRIMARY OUTCOMES:
Primary performance patient assessment | Change from Baseline in Constant Murley Score at 2-year post-op
  Constant Murley Score

CONTACTS AND LOCATIONS:
Overall Officials: Carrie Hill, Study Director — Conventus Orthopaedics, Inc.
Locations (5):
- United States (5):
  - Stanford University Hospital, Redwood City, California
  - Harbor-UCLA, Torrance, California
  - The Johns Hopkins University, Baltimore, Maryland
  - Snug Harbor Orthopedics, Duxbury, Massachusetts
  - Hennepin County Medical Center, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: Undecided